CLINICAL TRIAL: NCT00773630
Title: A Mono-center Study in Healthy Volunteers on the Comparative Bioavailability of Pletal 100 mg Tablets and a New Pletal 100 mg Orodispersible Tablet (ODT), This Latter in Fasting Conditions With and Without Water and Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Frankfurt Research Institute GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-08-101
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2009-03

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator): Intake of Pletal 100 mg tablets dose together with 200 ml water
  Interventions: Drug: Cilostazol
- B (Experimental): Intake of Pletal 100 mg ODT dose without water
  Interventions: Drug: Cilostazol
- C (Experimental): Intake of Pletal 100 mg ODT dose together with 200 ml water
  Interventions: Drug: Cilostazol
- D (Active Comparator): Intake of Pletal 100 mg ODT dose without water
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Cilostazol — 100 mg Cilostazol

SUMMARY:
The primary objective of this trial is to test whether Pletal ODT administered without water can be considered bioequivalent to Pletal administered with 200 ml water (both treatments being administered after fasting and at least 30 minutes prior to receiving a light breakfast) based on the standard pharmacokinetic variables.

The secondary objective is to assess the effect of water and the effect of food on the administration of Pletal ODT based on standard pharmacokinetic variables.

ELIGIBILITY:
Inclusion Criteria:

1. healthy male and female subjects of Caucasian race
2. able to read, to write and to fully understand German language
3. having given voluntary written informed consent before first invasive screening examination procedure
4. aged 18 to 45 years, inclusive
5. BMI of 18 - 28 kg/m2
6. good health as determined by medical history, physical examination, vital signs, electrocardiogram (ECG, serum/urine biochemistry and hematology)

Exclusion Criteria:

1. clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing) drug hypersensitivity
2. known hypersensitivity to one of the IMP substances
3. severe digestive disorder or surgery of the digestive tract (except for appen¬dectomy)
4. clinically relevant renal disorders (albuminuria, chronic infections)
5. clinically relevant hepatic disorders
6. clinically relevant respiratory disorders
7. clinically relevant cardiovascular disorders, especially any history of ventricular tachycardia, ventricular fibrillation or multifocal ventricular ectopics, or a history of additional risk factors for torsades de pointes (TdP) (e.g. heart failure, hypokalemia, congenital long QT-syndrome)
8. diabetes mellitus and thyroid dysfunction or other endocrine disorders
9. malignancy
10. substance abuse or addiction (alcohol, illicit drugs) in the past 3 years
11. neurologic or psychiatric illness
12. known predisposition to bleeding (e.g. active peptic ulceration, recent (within 6 month) haemorrhagic stroke, surgery within the previous three months, proliferative diabetic retinopathy, poorly controlled hypertension)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve, maximal concentration (Cmax) | 1-2 months

SECONDARY OUTCOMES:
Time of maximum (tmax), Vss/f, CL/f) | 1-2 months

CONTACTS AND LOCATIONS:
Overall Officials: Margarete Mueller, Dr., Principal Investigator — AAIPharma Deutschland GmbH & Co. KG
Locations (1):
- AAIPharma Deutschland GmbH & Co. KG, Neu-Ulm, Germany